CLINICAL TRIAL: NCT00582764
Title: Quantitative Dynamic Contrast Enhanced Breast MRI
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Oregon Health and Science University (Other); DeltaPoint,Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 05-091
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: Breast Lesion; Lesion; Breast; Cancer; 05-091
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — delta 24-sterol reductase; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Any patient undergoing MRI guided preoperative needle localization or MRI guided biopsy of the breast.
  Interventions: Other: perform dynamic contrast enhanced (DCE) MRI

INTERVENTIONS:
Other: perform dynamic contrast enhanced (DCE) MRI — With an IV catheter in place, the patient will lie prone on the MRI scanner table with the breasts positioned in the commercial breast coil and then be moved feet first to the center of the MRI scanner. The only difference introduced by the addition of DCE MRI is that before the patient is moved into the scanner for the first time, the IV catheter will be hooked up with a programmable power injector (Medrad, Indianola, PA) which is loaded with Gd contrast and saline. The contrast injection and saline flush will be delivered by the injector while the patient is inside the scanner and the DCE MRI data collection is in process. The Gd contrast dose used for DCE MRI is the same as for clinical MRI: 0.1 mmol/kg. The injection speed of 2 mL/sec is safe and similar to that of manual injection.

SUMMARY:
The purpose of this study is to see if dynamic contrast enhanced (DCE) MRI imaging makes it possible to distinguish benign conditions of the breast from malignant tumors and provide better information than can be obtained with regular MRI. DCE MRI uses a new way of collecting and analyzing the images or pictures which provides doctors extra information not available with standard imaging methods. This includes information about the blood vessels of different breast diseases. Pictures produced this way look just like the regular MRI pictures. The DCE MRI adds another imaging sequence (another scan) to the MRI examination ordered by your physician to evaluate your breast lesion, thus increasing the exam time (extra 10 min). The information gained from doing the new test, the DCE MRI, will not be used in your treatment and will not affect the type of care you receive for your breast lesions.

DETAILED DESCRIPTION:
Our aim is to perform dynamic contrast enhanced (DCE) MRI on 150 patients during their routine breast MRI examination at MSKCC. This will add extra 10 min scanning time to the routine examination. High resolution (submillimeter) parametric maps of pathophysiologic quantities, such as tumor vessel permeability, tumor perfusion, extracellular extravascular volume fraction, will be generated from the DCE MRI data. These results will be correlated with pathology to determine new pharmacokinetic threshold so that the negative predictive value for benign lesions is close to 100%. The improvement in diagnostic specificity may help to reduce unnecessary biopsies in the future.

ELIGIBILITY:
Inclusion Criteria:

· scheduled for breast MRI interventional procedure for a known breast lesion.

Exclusion Criteria:

* patients who would be normally excluded from undergoing an MRI examination patients with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field.
* patients who are unable to cooperate for an MRI, and/or have known reaction to gadolinium contrast agent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected at the time of the MRI interventional procedure by the radiologist who is protocoling the MRI examinations and who is an investigator on this protocol. Any known breast lesion, benign or malignant, will be appropriate for evaluation with DCE MRI. Pathology results will be obtained for each patient as a result of surgery or MRI guided biopsy, allowing correlation between the pathology and DCE MRI data.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2005-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To assess whether the new quantitative MRI method can discriminate between malignant and nonmalignant breast lesions among the lesions seen in conventional MRI. | December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Sunitha Thakur, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center website — http://www.mskcc.org